CLINICAL TRIAL: NCT06127017
Title: Comparing Marginal Bone Loss for Immediately Loaded Implants in Maxillary Full Arch Interim Prosthesis Using Welded Titanium Bar Versus Polyetheretherketone Bar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, soha saeid mohammed, Assistant lecturer, Oral and maxillofacial prosthodontics department, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1226
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Edentulous Jaw
Keywords: immediate loading, interim prosthesis, intra oral welding
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titanium bar (Placebo Comparator): 6 implants in each participant will be immediately loaded and splinted with intraorally welded titanium bar.
  Interventions: Procedure: splinting dental implants with titanium bar
- PEEK bar (Active Comparator): 6 implants in each participant will be immediately loaded and splinted with PEEK bar.
  Interventions: Procedure: splinting dental implants with PEEK bar

INTERVENTIONS:
Procedure: splinting dental implants with titanium bar — splinting of dental implants will be done in the placebo comparator group by welding a titanium bar intraorally to the temporary sleeves attached to the implants.
  Arms: Titanium bar
Procedure: splinting dental implants with PEEK bar — in the active comparator group ,the PEEK bar will be attached to the temporary sleeves using flowable composite resin material.
  Arms: PEEK bar

SUMMARY:
Fourteen completely edentulous patients will be randomly allocated into two parallel arm groups. For both groups virtual implant planning will be done and surgical guide will be planned and printed. An immediate interim full arch PMMA prosthesis will be virtually designed and printed for both groups. For the Intraoral welding group, seven patients will receive immediately loaded interim fixed full arch prosthesis splinted by intraoral welded bar. While for PEEK group in which seven patients will receive immediately loaded interim fixed full arch prosthesis splinted by PEEK bar. Marginal bone loss will be clinically evaluated at four, six months follow up period using CBCT.

DETAILED DESCRIPTION:
Study settings The study will be conducted in Oral & Maxillofacial Prosthodontics Department, Faculty of Dentistry, Ain Shams University. Sample size calculation Fourteen patients will be selected to share in this study from the outpatient clinic of Prosthodontics Department, Faculty of Dentistry, Ain-Shams University. G power program (3. 1) was used for calculations of sample size. Statistical calculator was based on 95% confidence interval and power of the study 80% with α error 5%.

Based on a previous study (Degidi, Marco, Diego Nardi, and Adriano Piattelli. "Prospective study with a 2-year follow-up on immediate implant loading in the edentulous mandible with a definitive restoration using intra-oral welding), which showed that the mean of marginal bone growth was 0.21 in one group compared to the second group. Using un paired t test the results were found to be significant. So, it was relied upon in this study. Based on this assumption, sample size was calculated according to these values producing a minimal sample size of fourteen patients being enough to find such a difference. Study procedures

1. Randomization and allocation concealment techniques Computer-generated random numbers will be used for simple randomization of the subjects. Therefore, the participants will be randomly allocated into two groups: intraoral welding group and PEEK group. The allocation ration will be set 1:1. Allocation concealment will be done using opaque sealed envelopes.
2. Details of intervention:

Ethical approval will be granted by the Research Ethical Committee, Faculty of Dentistry, Ain Shams University (FDASUREC). All patients will be informed in details about the nature of investigation and the aim of the study. Patient's data will be kept safe and confidential to protect the security and privacy of the patient information. All participants will be given notice about their privacy and their rights. 1-Patient Grouping: Fourteen patients will be enrolled in this study and randomly divided into two groups as follow Group Ⅰ: seven patients will receive immediately loaded interim fixed full arch prosthesis splinted by intraoral welded bar. Group Ⅱ: seven patients will receive immediately loaded interim fixed full arch prosthesis splinted by PEEK bar

2-Patient selection: The inclusion criteria will be systemically free completely edentulous patient ranged from 45 y to 69 years old with Class I maxillary-mandibular relationship, Normal salivary flow with normal viscosity. Residual maxillary ridge has adequate bone and covered by firm healthy mucosa. The excluded patients will include patients with major systemic diseases that may affect osseointegration as uncontrolled diabetes or under bisphosphonate treatment, Patients with poor oral hygiene. Patients with abnormal oral habits as (bruxism, clenching, tongue thrusting).Potentially uncooperative patients who are not willing to go through the proposed interventions. 3-Clinical steps:

a. pre-surgical procedures: i. Patients' history: Medical history: Patients will be asked about their medical and dental history through a direct interview and a detailed questionnaire sheet. Dental history: Patients will be asked about the cause, the date of teeth extraction and if there is any previous experience with any prosthetic appliance, any problems with TMJ will also be recorded. ii. Patients' examination:

Extra oral examination:

Extraoral examination will be performed for the detection of any abnormal facial anomalies, skin inflammation or lesions, any abnormalities in the TMJ as joint clicking, limitation in mouth opening or pain, and checking the maxillo-mandibular relationship Intra-oral examination: Visual and digital examination will be performed following routine procedures to examine denture bearing mucosa, border tissues, abnormal soft tissue, tongue, frenula, muscle tone, saliva, tori, sharp bony spicules, remaining teeth, arch relationship, ridge form, inter-ridge space and undercuts..

Radiographic evaluation:

(CBCT) radiograph will be done to evaluate the degree of bone resorption, quality and quantity of bone, to detect if there are remaining roots and any pathological lesions

Prosthetic procedures:

Properly constructed conventional single upper denture will be made for all patients. The Conventional denture will be duplicated with radiopaque markers and CBCT will be used to determine the exact positions of the implants. Virtual implant planning will be done using the BlueSky Bio 4 software. A surgical guide will be planned and then the 3D virtual guide will be exported as STL file to the 3D printing machine. An immediate interim full arch PMMA prosthesis will be virtually designed and printed for both groups. For the second group a PEEK bar will be virtually designed and printed. b. Surgical procedure: Surgery will be done under local anesthesia. The surgical guide will be fixed in place. Six implants will be placed according to the planned cone beam CT using surgical guide to accurately place the implants. Implants will be distributed following the Misch protocol; two implants in the first molar position, two implants in the canines position and two implants in the first centrals position. Serial osteotomies will be performed using sharp drills under copious irrigation to decrease heat generation until the planned depth and width will be reached.

The implant will be inserted through the osteotomy manually then continued using a ratchet with 35 Ncm torque Multiunit abutments will be screwed to the implants according to the Virtual implant planning. Titanium cylinders will be connected to the multiunit abutments.

Adjustment of the interim prosthesis and immediate loading:

All the pick-up procedures will be done in the same session of implant installation for both groups.

1. For the intraoral welding group:

   A titanium bar will be welded to titanium cylinders using an intraoral welding unit.

   Then, pick up will be done for the printed interim PMMA prosthesis to the titanium bar.
2. For the PEEK group:

The virtually designed and printed PEEK bar will be cemented to the titanium cylinders using flowable composite then, pick up will be done for the printed interim PMMA prosthesis to the printed PEEK bar. 4-Method of evaluation: Implant marginal bone loss (MBL) will be the difference in marginal bone level from the functional loading time with the interim prosthesis (T0) to the end of the follow-up (T1after four months, T2 after six months) .Marginal bone level around the implant will be measured from the CBCT scans made at T0, T1, T2. Vertical buccal or lingual bone heights (VBBH or VLBH) and horizontal buccal or lingual bone thicknesses (HBBT or HLBT) at the implant platform will be measured at themidsagittal cut of each implant perpendicular to the dental arch on the CBCT scan.

The distance from the implant platform (the horizontal interface between the abutment and the implant) to the most coronal point of bone-to-implant contact will be taken as the vertical bone height. Measurements will be calibrated by using the actual known length of the implant. Similarly, the vertical mesial or distal bone height (VMBH or VDBH) at the implant platform will be measured at the midsagittal cut of each implant parallel to the dental arch on the CBCT scan

ELIGIBILITY:
Inclusion Criteria:

.medically free. .class I maxillomandibular relation. .normal salivary flow.

* residual ridge has adequate mucosa
* covered with firm healthy mucosa.

Exclusion Criteria:

. poor oral hygiene. .uncooperative patients. .patients with abnormal oral habits.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
marginal bone loss measurement | total frame of 6 months with the following frequencies :at base line, after 4 months and after 6 months.
  marginal bone loss will be measured using cone beam computed tomography at the buccal, palatal, mesial and distal aspect of the implant and an average value will be calculated for each implant.

CONTACTS AND LOCATIONS:
Overall Officials: soha s elsaeid, Principal Investigator — Assistant lecturer ,Faculty of Dentistry, Ain Shams university

IPD SHARING:
Plan to Share IPD: No